CLINICAL TRIAL: NCT03470428
Title: Clinical Characteristics and Associations of the "Good Fontan" Patient
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: New England Congenital Cardiology Association (NECCA) (Unknown); Yale University (Other); Dartmouth College (Other); Connecticut Children's Medical Center (Other); University of Vermont (Other); Child Heart Associates (Unknown); Congenital Heart (Unknown); University of Massachusetts, Worcester (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rahul Rathod, Cardiologist, Boston Children's Hospital
Other Study IDs: IRB-P00024716
Record Dates: First submitted 2018-03-06; First posted 2018-03-20 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Disease; Single-ventricle
Keywords: Fontan; Single Ventricle
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric Fontan Patients: Participants ages 10 to 18 who have had Lateral Tunnel or Extracardiac Fontan procedures.
- Adult Fontan Patients: Participants ages 18 to 60 who have had Lateral Tunnel or Extracardiac Fontan procedures.

SUMMARY:
This study aims to determine what are some of the clinical characteristics and associations of Fontan patients who are doing well, as well as how accurate cardiology providers are at predicting the likelihood of future adverse event in their Fontan patients.

DETAILED DESCRIPTION:
This is a multi-center prospective study that involves collecting data from patients as well as their cardiology providers in order to determine whether there is correlation between patient-reported quality of life assessments and clinician-identified assessments of their patients. The study also involves collecting data from the medical records of participating patients and entering it into our study database.

ELIGIBILITY:
Inclusion Criteria:

* Extracardiac or Lateral Funnel Fontan

Exclusion Criteria:

* Currently being evaluated for or listed for cardiac transplant
* Underwent Fontan revision or conversion
* Currently pregnant

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with congenital heart disease who have undergone the Fontan procedure.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Surprise question | 1 year
  The ability of the cardiologist's response to the "surprise" question to predict adverse cardiac events within 1 year

SECONDARY OUTCOMES:
Clinical characteristics and associations of the "good Fontan" | 1 year
  Clinical characteristics and associations of this group (the "good Fontan") are different compared to those that are in the "at-risk" category (all others that do not fit into the "good Fontan" category). Data measurements will include relevant clinical data available for each patient, including but not limited to data from cardiac surgeries, catheterizations, MRIs, echocardiograms, exercise stress tests, current medications, labs, and patient responses to questionnaires.
Correlation between patient and provider assessments | 1 year
  There will be a positive correlation of the patient's own assessment of quality of life with the clinician-identified designation of a "good Fontan."
Clinician factors associated with adverse events conversation with patients | 1 year
  Clinician factors (years of experience, primary subspecialty, gender, parenthood) are associated with beliefs in regard to appropriate timing to discuss potential long-term adverse events to Fontan patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Rathod, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] d'Udekem Y, Iyengar AJ, Cochrane AD, Grigg LE, Ramsay JM, Wheaton GR, Penny DJ, Brizard CP. The Fontan procedure: contemporary techniques have improved long-term outcomes. Circulation. 2007 Sep 11;116(11 Suppl):I157-64. doi: 10.1161/CIRCULATIONAHA.106.676445. PMID 17846297
- [Background] Diller GP, Giardini A, Dimopoulos K, Gargiulo G, Muller J, Derrick G, Giannakoulas G, Khambadkone S, Lammers AE, Picchio FM, Gatzoulis MA, Hager A. Predictors of morbidity and mortality in contemporary Fontan patients: results from a multicenter study including cardiopulmonary exercise testing in 321 patients. Eur Heart J. 2010 Dec;31(24):3073-83. doi: 10.1093/eurheartj/ehq356. Epub 2010 Oct 7. PMID 20929979
- [Background] Blume ED, Balkin EM, Aiyagari R, Ziniel S, Beke DM, Thiagarajan R, Taylor L, Kulik T, Pituch K, Wolfe J. Parental perspectives on suffering and quality of life at end-of-life in children with advanced heart disease: an exploratory study*. Pediatr Crit Care Med. 2014 May;15(4):336-42. doi: 10.1097/PCC.0000000000000072. PMID 24583501
- [Background] Lakin JR, Robinson MG, Bernacki RE, Powers BW, Block SD, Cunningham R, Obermeyer Z. Estimating 1-Year Mortality for High-Risk Primary Care Patients Using the "Surprise" Question. JAMA Intern Med. 2016 Dec 1;176(12):1863-1865. doi: 10.1001/jamainternmed.2016.5928. No abstract available. PMID 27695853
- [Background] Hamano J, Morita T, Inoue S, Ikenaga M, Matsumoto Y, Sekine R, Yamaguchi T, Hirohashi T, Tajima T, Tatara R, Watanabe H, Otani H, Takigawa C, Matsuda Y, Nagaoka H, Mori M, Yamamoto N, Shimizu M, Sasara T, Kinoshita H. Surprise Questions for Survival Prediction in Patients With Advanced Cancer: A Multicenter Prospective Cohort Study. Oncologist. 2015 Jul;20(7):839-44. doi: 10.1634/theoncologist.2015-0015. Epub 2015 Jun 8. PMID 26054631